CLINICAL TRIAL: NCT05474846
Title: Combination Therapy for Treatment of Sleep Disturbance in Patients With Advanced Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0180; NCI-2022-06045 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Sleep; Fatigue; Anxiety; Cancer; Depression
MeSH Terms: conditions — Fatigue; Anxiety Disorders; Neoplasms; Depression | interventions — Melatonin; Cognitive Behavioral Therapy; Methylphenidate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Combination Therapy (BLT+MT+MP with CBT) (Experimental): Patients receive Melatonin (called MT) PO QD for 6 weeks, Methylphenidate (called MP) PO BID for 6 weeks, Bright Light Therapy (called BLT) for 30 minutes daily for 6 weeks, and Cognitive Behavior Therapy (called CBT) weekly for 6 weeks.
  Interventions: Drug: Melatonin; Other: Placebo for Melatonin; Drug: Methylphenidate
- Placebo (CLT+ placebo MT + placebo MP with CBT) (Experimental): Patients receive placebo Melatonin (called placebo MT) PO QD for 6 weeks, placebo Methylphenidate (called placebo MP) PO BID for 6 weeks, Control Light Therapy (called CLT) for 30 minutes daily for 6 weeks and Cognitive Behavior Therapy (called CBT) weekly for 6 weeks.
  Interventions: Drug: Melatonin; Other: Placebo for Melatonin
- Bright light and Melatonin (BLT + MT+ placebo MP with CBT) (Experimental): Patients receive Bright Light Therapy (called BLT) for 30 minutes daily for 6 weeks, Melatonin (called MT) PO QD for 6 weeks, placebo Methylphenidate (called placebo MP) PO BID for 6 weeks, and Cognitive Behavior Therapy (called CBT) weekly for 6 weeks.
  Interventions: Other: Placebo for Melatonin; Drug: Methylphenidate
- Methylphenidate (CLT + placebo MT + MP with CBT) (Experimental): Patients receive Control Light Therapy (called CLT) for 30 minutes daily for 6 weeks, placebo Melatonin (called placebo MT) PO QD for 6 weeks, Methylphenidate (called MP) PO BID for 6 weeks, and Cognitive Behavior Therapy (called CBT) weekly for 6 weeks.
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Given by PO
  Other Names: Methylphenidate Given by PO; Behavioral: Bright Light Therapy; Behavioral: Cognitive Behavior Therapy
  Arms: Combination Therapy (BLT+MT+MP with CBT); Placebo (CLT+ placebo MT + placebo MP with CBT)
Other: Placebo for Melatonin — Given by PO
  Other Names: Placebo for Methylphendate Given by PO; Control Light Therapy Sham Therapy; behavioral: Cognitive Behavior Therapy Counseling session
  Arms: Bright light and Melatonin (BLT + MT+ placebo MP with CBT); Combination Therapy (BLT+MT+MP with CBT); Placebo (CLT+ placebo MT + placebo MP with CBT)
Drug: Melatonin — Given by PO
  Other Names: Placebo for Methylphenidate Given by PO; Behavioral: Bright Light Therapy Given by PO; Behavioral: Cognitive Behavior Therapy Counseling session
  Arms: Combination Therapy (BLT+MT+MP with CBT); Methylphenidate (CLT + placebo MT + MP with CBT)
Drug: Methylphenidate — Given by PO
  Other Names: Placebo for Melatonin Given by PO; Control Light Therapy Sham Therapy; Behavioral: Cognitive Behavior Therapy Counseling session
  Arms: Bright light and Melatonin (BLT + MT+ placebo MP with CBT); Combination Therapy (BLT+MT+MP with CBT)

SUMMARY:
To learn if Cognitive Behavior Therapy (called CBT), combined with either Bright Light Therapy (called BLT), methylphenidate, and/or melatonin, can help improve sleep and other related symptoms such as fatigue, anxiety, and depression in cancer patients. This is an investigational study. In this study, BLT, Methylphenidate and Melatonin will be compared to their placebos.

DETAILED DESCRIPTION:
Objectives:

Primary:

To compare the effects of the combination therapy arm with the placebo arm on sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) at the end of 6 weeks (primary end point). We hypothesize that there will be a greater maintenance of sleep quality in the combination arm than in the placebo arm after 6 weeks.

Secondary:

To compare the effects of the combination therapy arm with the placebo arm on sleep quality (PSQI) at 3- and 6-months post-intervention. We hypothesize that there will be a greater maintenance of sleep quality in the combination arm than in the placebo arm at 3- and 6-months post intervention.

Secondary:

To compare the effects of the remaining active therapy arms with the placebo and combination arms on sleep quality (PSQI) at all post-intervention assessments. We hypothesize that there will be a greater maintenance of sleep quality in the active arms than in the placebo arm at all post-intervention assessments. Additionally, there will be greater maintenance of sleep quality in the combination arm than in the remaining active arms.

Secondary:

To compare the effects of the active therapy arm and the placebo arm for sleep-wake cycle disturbance (Actigraphy - sleep onset latency, wake after sleep onset, total sleep time, sleep efficiency, and mean daytime activity). We hypothesize that there w/ill be greater maintenance of sleep-wake cycle (synchronization) in the combination therapy arm.

Secondary:

To determine whether the addition of MP to BLT+MT synergistically maintains sleep quality as measured by change from baseline PSQI. We hypothesize that MP and BLT+MT will synergistically maintain sleep quality.

Exploratory:

To explore the effects of the active therapy arm on psychological symptoms (Hospital Anxiety and Depression Scale), fatigue (Functional Assessment of Chronic Illness Therapy - Fatigue), sleep and related symptoms (PROMIS-Sleep), inflammation (C-reactive protein), resting-state cognition (Amsterdam resting-state questionnaire, ARSQ) and quality of life (Functional Assessment of Cancer Therapy - General) and how they vary over time. We hypothesize that there will be more promotion of sleep related symptoms and quality of life in the combination therapy arm than in the placebo, BLT, and Methylphenidate arms.

Exploratory:

To explore changes in brain function and structure (using functional, structural and diffusion-weighted MRI) and changes in resting-state cognition (ARSQ) and sleep symptoms following (a) combination therapy arm (i.e., CBT + BLT + MP + MT); (b) CBT + BLT + MT + placebo (MP); (c) CBT + MP + placebo (control light + MT); and (d) CBT + placebo (control light + MT + MP). We hypothesize that in patients with advanced cancer and sleep disturbances, there will be changes in (a) resting-state brain connectivity within the default-mode network; (b) cortical volume within specific brain areas including bilateral thalamus; and (c) white-matter water diffusion in specific fibers tracts that underline directed functional connectivity, including connectivity between the pulvinar, agranular frontal area and the parietal cortex - following (a-d) therapy arms; and (e) improvements in brain function and structure will be the most robust in combination therapy arm than placebo arm. We further hypothesize that improvements in brain function and structure will be associated with improvements in resting-state cognition and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. presence of poor sleep quality, defined as Pittsburgh Sleep Quality Index (PSQI) total score ≥ 5, with patients describing poor sleep as being present for a minimum of 2 weeks;
2. ability to communicate in English;
3. cognitively competent to respond appropriately to questions, as measured by the Memorial Delirium Assessment Scale (MDAS) (≤ 13/30);
4. willing and able to sign a written informed consent;
5. life expectancy of ≥ 1 year as assessed by the oncologist or the principal investigator (SY) using the "surprise question," "Would I be surprised if this patient died in the next 12 months?"; and
6. no pain or stable pain (defined as pain ≤ 4 on Edmonton Symptom Assessment Scale (ESAS) or under control and on stable doses of opioids for 1 month).
7. Age 18 years or older
8. be willing to complete in-person or telemedicine follow-up visits with research staff, and able to complete CBT intervention either in person or virtually within Texas.

Exclusion Criteria:

1. active use of systemic anti-inflammatory prescription medications including steroids; unless used during or prior to cancer treatment as a prophylaxis (i.e., nausea);
2. known history of psychiatric illness (e.g., schizophrenia, bipolar disorder, major depressive disorder), sleep disorder (e.g., obstructive sleep apnea, narcolepsy, periodic limb movement disorder), obesity hypoventilation syndrome, glaucoma, congenital blindness, self-reported acquired blindness, significant cataracts or retinal disease; and night shift workers.
3. Hospital Anxiety and Depression (HADS) score ≥21, or use of antidepressants, unless the patient is receiving a stable dose for at least 1 month;
4. use of hypnosedative drugs or stimulants; unless on stable doses of hypnosedative drugs or stimulants for at least 1 month;
5. use of monoamine oxidase inhibitors (MOI), tricyclic anti-depressants and anticoagulants; and
6. patients who have bright sunlight exposure for consecutive 30 minutes or more daily in the past month, or prior exposure to BLT, or prior use of MT, MP, or CBT.
7. other medical reason that increases patient risk as determined by PI.
8. For patients participating in the MRI data collection component of the study, we will exclude the participants who meet the following criteria:

   1. . Any metallic objects in the body. Metal plates, certain types of dental braces, cardiac pacemakers, ext., that are sensitive to electromagnetic fields contraindicate MRI scans
   2. . Claustrophobia
9. Pregnancy as documented in the medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) questionnaires | Through the study completion, an average of 1 year.
  Pittsburgh Sleep Quality Index (PSQI) questionnaire score on a 4-point scale ranging from 0 (not during the 2 weeks) to 3 (3 or more times a week).

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, MD, Principal Investigator — MD Anderson
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org